CLINICAL TRIAL: NCT07334834
Title: Implementation of an Algorithm- and Multi-professional Team-supported Strategy to Improve Lipid Management of Patients With Atherosclerotic Cardiovascular Disease: OPTIMIZE ASCVD
Brief Title: Implementation of an Algorithm- and Multi-professional Team-supported Strategy to Improve Lipid Management of Patients With Atherosclerotic Cardiovascular Disease
Acronym: OPTIMIZE ASCVD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Prevention Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202401CPC
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hyperlipidemia
Keywords: Lipid Management; Atherosclerotic Cardiovascular Disease; Coronary Artery Disease; Peripheral Artery Disease; Carotid Artery Disease
MeSH Terms: conditions — Hyperlipidemias; Atherosclerosis; Coronary Artery Disease; Peripheral Arterial Disease; Carotid Artery Diseases | interventions — Algorithms

STUDY DESIGN:
Intervention Model Description: Comparative Effectiveness
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Guideline-directed lipid management by usual care provider (Other)
  Interventions: Other: Guideline-directed lipid management by usual care provider
- Algorithm- and multi-professional team-supported lipid management (Experimental)
  Interventions: Other: Algorithm- and multi-professional team-supported lipid management

INTERVENTIONS:
Other: Algorithm- and multi-professional team-supported lipid management — Algorithm- and multi-professional team-supported lipid management
  Other Names: Experimental
  Arms: Algorithm- and multi-professional team-supported lipid management
Other: Guideline-directed lipid management by usual care provider — Guideline-directed lipid management by usual care provider
  Other Names: Control
  Arms: Control: Guideline-directed lipid management by usual care provider

SUMMARY:
This is a randomized, controlled, collaborative, multicenter, pilot implementation science study evaluating the hypothesis that algorithm- and multi-professional team-supported lipid management reduces low density lipoprotein-cholesterol (LDL-C) compared with usual care in patients with atherosclerotic cardiovascular disease (ASCVD).

DETAILED DESCRIPTION:
OPTIMIZE-ASCVD is a randomized, controlled, collaborative, open-label, multicenter pilot implementation science study evaluating the hypothesis that algorithm- (Appendix A) and multi-professional team-supported lipid management reduces LDL-C compared with usual care in patients with ASCVD.

Approximately 100 participants will be randomized (1:1).

* Participant preference for injectable vs oral lipid therapy will be recorded at baseline.
* Participants allocated to algorithm-and multi-professional team-supported lipid management will be evaluated by a physician and prescribed lipid therapy which aims to achieve LDL-C target without titration. Participants will be contacted by a pharmacist to provide education about the medication and support any access issues.
* Participants allocated to usual care will be referred for management by their usual care provider who will receive a summary of guideline recommendations

The study will include decentralized clinical trial features including use of local, Clinical Laboratory Improvement Amendments (CLIA)-certified laboratories for blood tests, use of data extracted from the electronic medical record (EMR), electronic collection of patient-reported outcomes (PRO) and remote conduct of study activities. As an open label study with both strategy groups receiving GDMT, no Data and Safety Monitoring Committee will be convened. Study leadership will monitor aggregate data during the trial and may modify the sample size and/or cap enrollment of subgroups to ensure consistency with design assumptions.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent
* Age >18 years inclusive at screening
* Documented atherosclerotic vascular disease including:

  * Coronary artery disease (prior revascularization, myocardial infarction, imaging evidence of coronary atherosclerosis)
  * Peripheral artery disease (prior revascularization, amputation, ankle: brachial index (ABI) ≤ 0.90, imaging evidence of extra-coronary atherosclerosis)
  * Carotid artery disease (prior endarterectomy or stenting of the extracranial carotid artery or imaging evidence of carotid atherosclerosis)
  * Imaging evidence of atherosclerotic vascular disease in a non-coronary vascular bed (e.g. aorta, mesenteric, renal)
  * LDL-C >70mg/dL

Exclusion Criteria:

* Any reason that, in the opinion of the investigator, the patient would be unable to adhere to the protocol for the duration of the study (e.g. terminal diagnosis, metastatic cancer) or in whom participation might result in harm.
* Planned active titration of current lipid-lowering therapy
* Myocardial infarction or arterial revascularization within prior 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The between group difference in LDL-C percent change | Baseline to 3 months

SECONDARY OUTCOMES:
Between group difference | Baseline to 1 and 6 months
  LDL-C percent change
Between group difference | 1, 3 and 6 months
  The proportion achieving LDL-C <55 mg/dL
Between group difference | 1, 3 and 6 months
  Proportion receiving combination lipid lowering Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bonaca, MD, Principal Investigator — Colorado Prevention Center
Locations (1):
- University of Colorado Health System (UCHealth), Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No